CLINICAL TRIAL: NCT02831075
Title: A Clinical Study Using Adipose-derived Stem Cells for Diabetic Foot
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jie Shen (Other Government)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Academy Military Medical Science, China (Industry); The Fifth Affiliated Hospital of Southern Medical University (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor-Investigator, Jie Shen, professor, The Third Affiliated Hospital of Southern Medical University
Organization: The Third Affiliated Hospital of Southern Medical University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Southern Medical University
Record Dates: First submitted 2016-07-09; First posted 2016-07-13 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Peripheral Vascular Disease; Ischemia; Diabetic Foot
Keywords: Adipose-derived Stem Cells
MeSH Terms: conditions — Peripheral Vascular Diseases; Ischemia; Diabetic Foot | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adipose-derived stem cell (Experimental): Mesenchymal stem cells derived from adipocyte transplantation
  Interventions: Biological: Adipose-derived stem cell
- saline (Placebo Comparator): saline injections
  Interventions: Biological: saline

INTERVENTIONS:
Biological: Adipose-derived stem cell — stem cell acquisition, processing and reinfection, to evaluate the efficacy of adipose-derived stem cell.
  Arms: Adipose-derived stem cell
Biological: saline
  Arms: saline

SUMMARY:
Stem cell therapy has been a new and effective therapy in recent years for diabetic foot.This study intends to establish an optimal clinical research program, and attempts to break the technical bottleneck in the stem cell therapy for treating diabetes related vascular complications.

DETAILED DESCRIPTION:
Diabetic foot is one of the most serious chronic complications of diabetic patients, and still lacking effective treatments.

Stem cell therapy has been a new and effective therapy in recent years for diabetic foot. Combined with the previous studies of our research group, this study intends to transform part of the results of this research, establish an optimal clinical research program, and attempts to break the technical bottleneck in the stem cell therapy for treating diabetes related vascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus Type 2 or Type 1
* Age between 18-80 years
* Chronic foot ulcer more than 6 weeks
* No sufficient response to best standard care delivered for six weeks.
* PAD up to Fontaine stage III or IV period
* CLI with the ankle brachial index (index ankle-brachial, ABI) <0.7 and (or) the -percutaneous oxygen partial pressure (oxygen tension transcutaneous, TcPO2) <30mmHg

Exclusion Criteria:

* HbA1c >12%
* Hemoglobin <10 mg/dl
* Creatinine clearance rate <30ml/min
* Systemic bacterial, viral infections (Mei Du, hepatitis, cytomegalovirus infection, - HIV, B19 infection, herpes virus infection) and sepsis
* Have accepted the treatment of stem cells or growth factors
* Have a history of malignant disease
* Pregnancy
* Mental illness history
* Abnormal coagulation function
* Allergic reaction
* Severe cardiac insufficiency (III-IV NYHA)
* Using vasoactive substances

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Area of diabetic foot ulcers | 3 months
  To determine the ability of MSC to facilitate and accelerate diabetic foot ulcers healing.

SECONDARY OUTCOMES:
Improvement of transcutaneous oxygen partial pressure (TcPO2) | 3 months
  Improvement of local perfusion.
Improvement of microvascular cutaneous reactivity by laser Doppler perfusion monitoring (LDPM) | 3 months
Pain (Visual-Analog Scale) | 3 months
  Measure of the subjective symptom of pain.
Walking distance (treadmill) if possible | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Shen, Principal Investigator — The Third Affiliated Hospital of Southern Medical University
Locations (1):
- the Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided